CLINICAL TRIAL: NCT06561659
Title: Testing a Brief Exercise Intervention in Hoarding Disorder
Acronym: Exercise BDNF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Hannah Levy, Staff Psychologist, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Masking Description: Participants and investigators will not know the condition assignment until the intervention is about to begin. So the informed consent process, the study eligibility interview, and the self-report measures will be completed prior to condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Condition (Active Comparator): For participants randomized to the exercise intervention, they will complete 30 minutes of brisk walking around the campus. They will be asked to maintain at least a moderate level of exercise intensity throughout the 30-minute walk.
  Interventions: Behavioral: Exercise Condition
- Relaxation Control Condition (Other): For participants randomized to the control group, they will sit in the testing room and watch informational videos about animals.
  Interventions: Behavioral: Relaxation Control Condition

INTERVENTIONS:
Behavioral: Exercise Condition — Already described in the arm description
  Arms: Exercise Condition
Behavioral: Relaxation Control Condition — Already described in the arm description
  Arms: Relaxation Control Condition

SUMMARY:
Hoarding disorder (HD) is characterized by difficulty discarding personal possessions due to significant emotional distress when parting with personal items. This leads to the accumulation of excessive clutter which compromises the normal use of living spaces. In addition to emotional distress, individuals with HD experience significant impairment in physical health. One study found an 11-fold increase in stroke risk, a 10-fold increase in cancer risk, and a 7-fold increase in cardiovascular disease in individuals with HD relative to a general population comparison group. Patients with HD are also more likely to experience obesity and metabolic diseases such as diabetes. The short-term goal of the proposed study is to determine whether a brief exercise intervention improves discarding-related distress and brain-derived neurotropic factor (BDNF) in individuals with HD relative to a relaxation control condition. Preliminary evidence suggests that BDNF may be associated with greater body mass index and more severe HD symptoms in patients with HD. BDNF is a well-studied growth factor which is involved in neuronal transmission, plasticity, and survival of many neuron systems that have been implicated in psychiatric disorders, including serotonin, glutamate, and dopamine. BDNF has been proposed as a mechanism of exercise interventions for psychiatric disorders, as even one session of exercise has been shown to increase BDNF levels. This study represents an initial first step towards the long-term goal of improving current treatments for HD. This is important because although current cognitive-behavioral treatments (CBT) are effective, only 35% of patients who receive these treatments actually benefit from them. In the proposed pilot study, the investigators will test whether 30 minutes of moderate-intensity exercise reduces the distress associated with discarding and increases BDNF levels in individuals with HD relative to a relaxation control. The investigators will recruit 22 individuals with a primary diagnosis of HD. They will be randomly assigned to exercise or control. Following the intervention, the investigators will assess BDNF via serum. Participants will complete a standardized discarding task which consists of sorting and discarding personal possessions. The central hypothesis is that those in the exercise condition will demonstrate lower distress during the discarding task and greater BDNF levels as compared to those in the relaxation control condition. Should the hypothesis be confirmed, the investigators will be well poised to conduct large-scale clinical trials testing exercise interventions as adjunctive or alternative treatments to standard CBT.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of hoarding disorder
* Age 45-65 years

Exclusion Criteria:

* Contraindications to engaging in exercise, including cardiovascular, metabolic, or renal disease, thyroid problems, uncontrolled hypertension
* Significant mobility issues that would preclude brisk walking
* Schizophrenia, bipolar disorder, serious suicidal risk, active substance use disorder, and cognitive impairment that may preclude the ability to provide informed consent and/or participate in study procedures

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale | Immediately before and immediately after discarding task
  Participants will be asked to rate their distress before and after the discarding task using the Subjective Units of Distress Scale (SUDS; 0 = no distress and 100 = worst distress imaginable).
Brain Derived Neurotropic Factor (BDNF) | Immediately after the intervention or control condition
  Serum BDNF

SECONDARY OUTCOMES:
Number of items discarded | Experimenter will tally the number of items kept vs. discarded immediately after the discarding task
  The number of items discarded vs. kept during the discarding task will be compared between conditions

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Levy, PhD, Principal Investigator — Hartford Hospital
Locations (1):
- Anxiety Disorders Center, Institute of Living, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No